CLINICAL TRIAL: NCT05840900
Title: Mindfulness, Optimism, and Resilience for Perinatal Health and Equity Study
Acronym: MORPHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nina Ayala (Other)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Sponsor-Investigator, Nina Ayala, Attending Physician, Maternal-Fetal Medicine, Women and Infants Hospital of Rhode Island
Organization: Women and Infants Hospital of Rhode Island (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1983168
Record Dates: First submitted 2023-04-17; First posted 2023-05-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Psychiatric Disorders
Keywords: dispositional optimism; mindfulness; adverse perinatal outcomes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and clinicians will not be blinded, but the outcomes assessor and analytic teams will be blinded to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-based mindfulness training (Experimental): App-based daily mindfulness training Standard prenatal and pregnancy care
  Interventions: Behavioral: Digital Mindfulness Training
- Usual Care (No Intervention): Standard prenatal and pregnancy care

INTERVENTIONS:
Behavioral: Digital Mindfulness Training — Once daily, 5-10 minute mindfulness exercises for 8 week intervention period using the existing perinatal mindfulness application Expectful
  Arms: App-based mindfulness training

SUMMARY:
Dispositional optimism (the general assumption that more good things than bad will occur across various life domains) has been tied to improved somatic and mental health outcomes. Dispositional optimism is malleable, although prior interventions have been time and resource intensive and thus are not well-tailored to the peripartum period. The purpose of this pilot study is to evaluate the feasibility and acceptability of a pregnancy-oriented mindfulness phone application (Expectful) versus standard care among first-time mothers with low dispositional optimism in early pregnancy. Other aims include evaluating the impact of Expectful use on dispositional optimism, adverse pregnancy outcomes (cesarean delivery, hypertensive disorders of pregnancy, and gestational diabetes) and postpartum post-traumatic stress symptoms.

DETAILED DESCRIPTION:
This randomized clinical trial of nulliparous women with low dispositional optimism in early pregnancy seeks to determine whether use of a pregnancy-oriented digital mindfulness application will be feasible and acceptable and show preliminary evidence of efficacy in improving dispositional optimism, reducing adverse perinatal outcomes and improving postpartum post-traumatic stress symptoms.

This pilot will include 100 women recruited from the obstetrical service at Women and Infants Hospital of Rhode Island. Women will be included if they are nulliparous, have a singleton pregnancy at <20 weeks gestational age, speak English and have low dispositional optimism (a score of ≤14 on the validated, Revised Life Orientation Test). Eligible participants will be randomized to either using the digital app Expectful or standard pregnancy care.

Women will be randomized with equal probability to the intervention group using block randomization stratified by race/ethnicity (Hispanic, non-Hispanic White/Other or non-Hispanic Black).

Women in the mindfulness training arm will complete 8 weeks of daily mindfulness training exercises using Expectful. Women in the standard care group will receive standard pregnancy and postpartum care. Pregnancy and labor management will be at the discretion of each participant's obstetric provider.

Participants in both groups will be asked to complete 4 questionnaires: one at enrollment, a post-intervention one at 8 weeks, at the time of delivery and at 6-8 weeks postpartum. Half of the participants in each arm (total n=50), will be asked to complete a qualitative, semi-structured interview on the role of optimism and other resilience factors in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* English speaking
* Nulliparous (no prior delivery at or greater than 20w0d gestation)
* Pregnant with singleton fetus
* <20w0d gestation
* Low dispositional optimism (score </= 14 on the Revised Life Orientation Test)
* Owns a smart phone

Exclusion Criteria:

* Plan to deliver at another institution
* Ongoing (≥1/week) mind-body practice including mindfulness training, meditation or yoga
* Pre-gestational hypertensive disorder
* Pre-gestational diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants completing the assigned mindfulness exercises | 8-week intervention period
  The intervention will be considered feasible if ≥75% participants complete >50% of the assigned daily mindfulness exercises over the 8-week intervention period
Intervention acceptability | After 8 week intervention period, approximately 16-28 weeks gestation.
  The intervention will be considered acceptable if ≥75% report "satisfied" or "very satisfied" on a post-intervention consumer satisfaction survey with a 5-point Likert scale from very unsatisfied to very satisfied.

SECONDARY OUTCOMES:
Dispositional optimism | Study enrollment and 6-12 weeks postpartum
  Change in dispositional optimism score (on validated Revised Life Orientation Test, scale range 0-24, higher scores indicate higher optimism) between enrollment and postpartum assessments
Cesarean delivery | Delivery
  Binary yes/no
Hypertensive disorder of pregnancy | 6-12 weeks postpartum
  Binary yes/no; includes gestational hypertension, pre-eclampsia with or without severe features, HELLP syndrome or eclampsia
Gestational diabetes mellitus | Delivery
  Binary yes/no
Preterm birth | Delivery
  Binary yes/no; Delivery between 20w0d and 36w6d gestation
Traumatic birth | Delivery
  Binary yes/no; Self-reported experience of birth as traumatic given concern for life or well-being of self or infant
Postpartum post-traumatic stress symptoms | 6-12 weeks postpartum
  Continuous scale score using the PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders (PCL-5, scale range 0-80, higher scores indicate worse post-traumatic stress symptoms)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Obstetrics and Gynecology Care Center, Providence, Rhode Island
  - Prenatal Diagnosis Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang E, Lewkowitz AK, Unger JA, Garfield CF, Miller ES. Smartphone Applications to Support Perinatal Mental Health. Obstet Gynecol. 2026 Feb 1;147(2):229-238. doi: 10.1097/AOG.0000000000006139. Epub 2025 Dec 18. PMID 41411652